CLINICAL TRIAL: NCT06756776
Title: Effects of Dry Needling Versus Stretching of Hamstrings Muscles With Lumber Sustained Natural Apophyseal Glides on Pain, Range of Motion, Muscle Length and Disability in Patients With Non-specific Low Back Pain
Brief Title: Dry Needling vs. Stretching for Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Misbah Sohail
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Non Specific Low Back Pain
Keywords: non-specific low back pain; dry needling; SNAGs; ROM; disability; muscle length
MeSH Terms: interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SNAGs on the lumbar spine and stretching (Experimental): Sustained Natural Apophyseal Glides (SNAGs) on the lumbar spine and stretching of the hamstring muscles will be administered to Group A.
  Interventions: Device: Hot pack; Other: Sustained Natural Apophyseal Glides (SNAG); Other: Passive Hamstring (HM) stretching; Device: Transcutaneous Electrical Nerve Stimulation
- SNAGs on the lumbar spine and dry needling (Active Comparator): Sustained Natural Apophyseal Glides (SNAGs) on the lumbar spine and dry needling on the hamstring muscles will be administered to Group B.
  Interventions: Device: Hot pack; Other: Sustained Natural Apophyseal Glides (SNAG); Other: Dry needling; Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Hot pack — The Hot Pack is a therapeutic intervention device designed to deliver localized heat to targeted areas of the body for a duration of 15 minutes. It provides deep, soothing heat that helps to relax muscles, increase blood circulation, and reduce pain and stiffness. The device is typically used to treat conditions such as muscle tension, joint pain, and chronic discomfort. By applying consistent heat, the Hot Pack promotes improved tissue flexibility and alleviates muscle spasms. It is user-friendly, ensuring safe and effective use when applied to affected areas, with adjustable heat settings to accommodate individual needs.
Other: Sustained Natural Apophyseal Glides (SNAG) — The Mulligan Sustained Natural Apophyseal Glides (SNAG) technique for the lumbar spine will be applied to participants in both groups. Participants will assume a stride standing position. The therapist will stand behind the participant as described by Mulligan, supporting the patient during the application of the technique and ensuring the required movement can be performed easily. The therapist will apply the mobilizing force parallel to the facet joint plane (in the cephalic direction) over the spinous processes of the respective symptomatic spinal levels in a sustained manner while the patient performs trunk flexion. The flexion position will be maintained for a few seconds, after which the participant will return to the starting position, with the therapist continuing to maintain the mobilizing force. Three sets of six repetitions will be performed on each symptomatic lumbar spinal level.
Other: Passive Hamstring (HM) stretching — Passive Hamstring (HM) stretching will be performed by a physical therapist experienced in the treatment of chronic low back pain (CLBP) and trained in the study protocol. The procedure will follow manual therapy stretching standards [22]. First, the physical therapist will explain the procedure to the participant and reassure them that the stretching can be stopped if it becomes too difficult to tolerate. With the participant lying supine, the stretched limb will be placed in maximal, pain-free hip flexion with the knee flexed. The physical therapist will then slowly and gradually extend the knee to the maximal pain-free position. In this position, participants should feel an intense stretching sensation in the back of the thigh. If this position causes pain in the lower back, the hip flexion will be reduced to the maximal, pain-free range of motion (ROM). A stopwatch will be used to ensure that the final position is held for 1 minute for each limb.
  Arms: Group A: SNAGs on the lumbar spine and stretching
Other: Dry needling — Subjects will be positioned prone on a treatment table with their feet over the edge of the table. Dry needling (DN) will be applied to the hamstring muscles at three locations, each for 1 minute, using a fast in-out, cone-shaped technique.
  Subjects will receive DN three times a week. To standardize the approach and optimize the application of DN, the points will be located approximately close to the motor points of the hamstring muscles.
  Two of the locations are in the long and short heads of the biceps femoris, at points located at 30% and 60% of a straight line from the ischial tuberosity to the fibular head. For the semitendinosus and semitendinosus muscles, the DN location will be selected at 60% of a straight line from the ischial tuberosity to the medial femoral epicondyle.
  Disposable sterilized stainless steel needles (0.3×60 mm; DongBang AcuPrime Ltd, Korea) will be used.
  Arms: SNAGs on the lumbar spine and dry needling
Device: Transcutaneous Electrical Nerve Stimulation — The TENS (Transcutaneous Electrical Nerve Stimulation) unit is a therapeutic device designed to alleviate pain through the use of electrical impulses. It works by delivering low-voltage electrical currents via electrodes placed on the skin, targeting the affected area. These electrical pulses help to block pain signals sent to the brain and stimulate the production of endorphins, the body's natural pain relievers. The TENS unit is commonly used for managing both acute and chronic pain conditions, including muscle pain, joint pain, and nerve-related discomfort. The device is adjustable, allowing users to customize the intensity, duration, and frequency of the electrical stimulation to meet their individual needs. It is non-invasive, easy to use, and can be applied at home or in clinical settings for effective pain management.

SUMMARY:
Chronic low back pain (CLBP) is one of the common health issues and a leading cause of reduced mobility. It is characterized by pain during functional activities and is often associated with hamstring tightness. CLBP affects individuals across all age groups. Various methods are used to address low back pain, including manual therapy. Manual therapy techniques include Maitland mobilizations, Kaltenborn mobilizations, Mulligan techniques, stretching, and others.

Several stretching techniques have been proposed, including static stretching, dynamic stretching, ballistic stretching, and proprioceptive neuromuscular facilitation (PNF). Among these, static and dynamic stretching are the most commonly used methods. Static stretching is considered one of the safest and easiest techniques, which can be performed passively or actively. Literature supports that stretching improves muscle flexibility, provides relaxation, reduces pain, and increases the range of motion (ROM).

Dry needling is another physical intervention technique that has been utilized for patients with musculoskeletal disorders. Current literature supports the use of dry needling for trigger points in hamstring muscles, which is a contributing factor to low back pain.

The objective of this study is to compare the effects of dry needling and stretching combined with sustained natural apophyseal glides (SNAGs) on pain, ROM, muscle length, and disability in patients with non-specific low back pain.

A randomized clinical trial will be conducted at Hijaz Hospital using convenience sampling to recruit participants. Patients will be allocated into two groups (Group A and Group B) through simple random sampling using sealed opaque envelopes. After conventional treatment, Group A will receive SNAGs and stretching, while Group B will receive SNAGs and dry needling.

Outcome measures will include the goniometer for ROM, the Modified Oswestry Disability Index (MODI) for disability, the Numeric Pain Rating Scale (NPRS) for pain, and the Finger-to-Floor Distance Test for hamstring flexibility. These measures will be assessed at baseline, at the 2nd week, and after 4 weeks. Data will be analyzed using SPSS software (version 21).

The normality of the data will be assessed using the Shapiro-Wilk test. Based on the results, parametric or non-parametric tests will be used for within-group and between-group comparisons. SNAGs and dry needling will be evaluated for their effectiveness in treating non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* minimum 3 months chronicity of low back pain
* with tight hamstrings and positive passive knee extension test (12)

Exclusion Criteria:

* Chronic systemic bony and soft tissue diseases
* Recent history of trauma
* Degenerative joint diseases
* Psychiatrist diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | baseline, 2 weeks, and 4 weeks
  The patient's level of pain will be assessed using the Numeric Pain Rating Scale (NPRS), which ranges from 0 to 10. A score of 0 indicates "no pain," while a score of 10 represents the "worst pain imaginable." (19)

SECONDARY OUTCOMES:
Fingertip to Floor distance test | baseline, 2 weeks, and 4 weeks
  The finger-to-floor distance test can be used to assess spine stiffness and evaluate the effects of exercise on spine stiffness in individuals with spine disorders, such as ankylosing spondylitis and back pain. The reliability of the fingertip-to-floor test in patients with low back pain (LBP), assessed using the Intraclass Correlation Coefficient (ICC) and the Bland-Altman method, is excellent. After a functional restoration program, which includes daily exercises for flexibility, the test demonstrated good sensitivity to change, with an effect size of 0.87 and a Standardized Response Mean (SRM) of 0.97. The interobserver reliability of the fingertip-to-floor test is also high, with an ICC of 0.97 (unpublished data).
Passive knee extension test | baseline, 2 weeks, and 4 weeks
  A study shows that the goniometer is reliable for measuring knee and elbow joint angles, with reliability values ranging from r = 0.67 to 0.70 (16). The purpose of the Passive Knee Extension Test (also known as the 90-90 Straight Leg Raise [SLR] hamstring test) is to assess the joint range of motion and the quality of its movement, particularly the 'end feel' of the joint. This test is commonly used to measure hamstring muscle tightness. A test-retest reliability study for this assessment shows a reliability range of 0.87 to 0.94, indicating high intra-rater reliability (21).
Modified Oswestry Disability Index (ODI) (Urdu version) | baseline, 2 weeks, and 4 weeks
  The Modified Oswestry Disability Index (ODI) (Urdu version) will be used to assess the patient's functional disability due to chronic low back pain at baseline (0 weeks) and after 4 weeks. The modified ODI has a reliability score of 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Hijaz Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No